CLINICAL TRIAL: NCT05309733
Title: A Long-term Follow-up Study of Patients Who Received VOR33
Status: Terminated | Type: Observational
Why Stopped: Lack of Funding
Sponsor: Vor Biopharma (Industry)
Responsible Party: Sponsor
Other Study IDs: VBP201
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AML; Acute Myeloid Leukemia; CD33; allogeneic; HCT; hematopoietic stem cell transplant; leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Cohort 1: All patients who have received any part of or all of a VOR33 genome-edited hematopoietic stem and progenitor cell therapy product.
  Interventions: Genetic: VOR33

INTERVENTIONS:
Genetic: VOR33 — VOR33 is an allogeneic CRISPR/Cas9 genome-edited hematopoietic stem and progenitor cell therapy product that lacks the CD33 myeloid protein.

SUMMARY:
VOR33 long-term follow-up (LTFU) study

DETAILED DESCRIPTION:
VBP201 study is the VOR33 long-term follow-up (LTFU) study focusing on assessing long term safety and efficacy of VOR33. This study may last up to 15 years (counted from the date of VOR33 infusion completion). All patients who have participated in a study involving the drug product VOR33 and have completed the applicable study or prematurely discontinued, but have at least received the VOR33 infusion, will be asked to participate in the LTFU study.

ELIGIBILITY:
Inclusion Criteria:

* A patient is included in this study if he/she:

  1. Has received any part of or all of a VOR33 infusion

Exclusion Criteria:

* There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have received any part of or all of a VOR33 genome-edited hematopoietic stem and progenitor cell therapy product.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Long term safety of VOR33 in patients who participated in a VOR33 study in terms of study product-related Adverse Events/Serious Adverse Events (AEs/SAEs). | Years 1-15
  Incidence of VOR33-related AEs/SAEs or deaths.

SECONDARY OUTCOMES:
Long term efficacy of VOR33 in patients who participated in a VOR33 study in terms of persistence of CD33-negative hematopoiesis, overall survival (OS), and monthly relapse free survival (RFS). | Years 1-15
  Percentage of CD33-negative hematopoiesis and change over time. Overall rates of RFS measured from the time of hematopoietic cell transplantation (HCT) to the date of disease relapse, and OS rates defined as the time from HCT to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Miami Cancer Institute, Miami, Florida
  - National Institutes of Health, Clinical Center, Bethesda, Maryland
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No